CLINICAL TRIAL: NCT02267083
Title: Phase 2 Efficacy and Safety Study of Intravenous GPX-150, an Anthracycline Analog, in Patients With Soft Tissue Sarcoma
Brief Title: Efficacy and Safety Study of GPX-150 to Treat Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gem Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPX-150-002
Record Dates: First submitted 2014-09-23; First posted 2014-10-17 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — 5-imino-13-deoxydoxorubicin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GPX-150 (Experimental): GPX-150 for Injection, 265 mg/m2, every 21 days for 16 cycles or until death, disease progression, or unacceptable toxicity, or subject withdrawal.
  Interventions: Drug: GPX-150 for Injection

INTERVENTIONS:
Drug: GPX-150 for Injection — GPX-150 at a starting dose of 265 mg/m2 every 21 days for 16 cycles or until death, disease progression, or unacceptable toxicity. The dose of GPX-150 may be reduced by 25% if any dose reduction criteria are met. Two reductions are allowed per subject during the course of the study.
  Other Names: GPX-150; 5-imino-13-deoxy-doxorubicin HCl

SUMMARY:
This study will assess the safety and efficacy of GPX-150 administered intravenously every 3 weeks in the treatment of patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
This is an open-label, single arm study of GPX-150 in patients with soft tissue sarcoma. Approximately 22 patients will be treated in this study. The population for this study is adult patients with histologically proven advanced and/or metastatic malignant soft tissue sarcoma of intermediate or high histologic grade.

All patients who meet all entry criteria will receive GPX-150 at a starting dose of 265 mg/m2 every 21 days for 16 cycles or until death, disease progression, or unacceptable toxicity or subject withdrawal.

Prior to initiation of treatment, subjects will undergo screening and baseline evaluations. During all study visits, subjects will be evaluated for safety. The dose of GPX-150 may be reduced when subjects meet specified dose reduction safety criteria. Subjects will be evaluated regularly for safety and tolerability. Tumor measurements will be calculated at baseline (within 28 days prior to treatment initiation), then at regular intervals while receiving treatment for up to 1 year. After discontinuing the treatment phase of the study, safety assessments and tumor measurements will be performed 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histological documentation of soft tissue sarcoma (biopsy may be historical and may have been obtained from primary tumor or a metastatic site).
3. Advanced and/or metastatic malignant soft tissue sarcoma of intermediate or high histologic grade. Excluded are the following sarcoma subtypes:

   * Well-differentiated liposarcoma or atypical lipomatous tumor
   * Embryonal or alveolar rhabdomyosarcoma
   * Ewing sarcoma of soft tissue or bone
   * Gastrointestinal stromal tumor (GIST)
   * Dermatofibrosarcoma protuberans
   * Alveolar soft part sarcoma
   * Solitary fibrous tumor
   * Clear cell sarcoma
   * Kaposi sarcoma
   * Extraskeletal myxoid chondrosarcoma
   * PEComa (perivascular epithelial cell tumor)
   * Myoepithelioma / mixed tumor
4. Measurable disease as per RECIST 1.1.
5. Subject has received either:

   * No prior chemotherapy for current sarcoma, or
   * A single course of gemcitabine and/or docetaxel as adjuvant therapy that was completed at least 6 months prior to planned first dose
6. ECOG Performance Status of 0 - 2.
7. Adequate cardiac function:

   * LVEF above the institution's lower limit of normal
   * QTcF ≤ 450 msec for males or 470 msec for females.
8. Willing and able to provide written informed consent.
9. Male and female subjects must agree to use a highly reliable method of birth control for the duration of the study.
10. Women of childbearing potential must have a serum pregnancy test performed within 28 days prior to the first day of study drug dosing.

Exclusion Criteria:

1. Sarcomas arising from bone or cartilage, e.g. chondrosarcoma, osteosarcoma, chordoma.
2. Subject is eligible for a potentially curative therapy.
3. Prior primary chemotherapy.
4. Prior radiotherapy to > 25% of bone marrow volume.
5. Treatment within 28 days prior to Dose 1 with:

   * Palliative surgery or radiotherapy.
   * Approved anticancer therapy including chemotherapy or immunotherapy.
   * Contraindicated treatments noted in the product labelling for doxorubicin, including trastuzumab and inhibitors and inducers of CYP3A4, CYP2D6, or P-gp.
   * An investigational therapy.
   * Any major surgery (e.g. requiring general anesthesia).
6. Inadequate bone marrow, liver, and renal function, as assessed by the following laboratory parameters:

   1. Absolute neutrophil count (ANC) < 1,500/mm3.
   2. Platelet count < 100,000/mm3.
   3. Total bilirubin > 1.5×ULN (upper limit of normal).
   4. ALT and AST > 2.5×ULN. For patients with documented liver metastases, ALT and AST > 5×ULN.
   5. Serum creatinine > 1.5 x ULN.
   6. International Normalized Ratio (INR) and activated partial thromboplastin time [PTT] ≥ 1.5×ULN, if not therapeutically anticoagulated.
   7. Serum albumin < 3.0 gm/dL.
7. Congestive heart failure > Class II New York Heart Association Functional Classification, current pericarditis, myocardial infarction within 6 months, or symptomatic coronary artery disease.
8. Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a patient and/or their compliance with the protocol.
9. Active infection requiring systemic antibacterial/antibiotic, antifungal, or antiviral therapy.
10. Documented metastases to brain or meninges.
11. Any malignancy other than soft tissue sarcoma within the last 5 years prior to screening, with the exception of cervical carcinoma in situ, basal cell carcinoma, or superficial bladder tumors that have been successfully and curatively treated with no evidence of recurrent or residual disease.
12. Body surface area (BSA) ≥ 2.4 m2.
13. Currently pregnant or nursing.
14. Known allergy to any of the study drugs or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01-07; Primary Completion 2015-11-11 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa Holden Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - University of Iowa Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GPX-150
Started | 22
Completed | 3
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: The Safety Population consists of all subjects who received at least 1 dose of GPX-150 and the Intent-to-Treat (ITT) Population consists of all subjects in the Safety Population who had at least one tumor assessment using RECIST 1.1 or who died prior to any tumor assessment.
Arm/Group | GPX-150
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Region of Enrollment [Number; unit: participants] — Subjects diagnosed with advanced and/or metastatic soft tissue sarcoma of intermediate or high histologic grade.
  participants
    United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Progression-free at 12 Months Per RECIST 1.1
Description: The primary efficacy endpoint is the number of patients who were progression-free at 12 months, which is obtained by inversion of the Kaplan-Meier curve for progression-free survival (PFS) at 12 months. Of note, the statistical comparison to historical sarcoma data described in the protocol was not performed due to an enrollment of less than the planned sample size of 30 subjects. Progression is defined using RECIST 1.1, as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: 12 months from the beginning of study treatment
Population: Consists of all subjects in the safety population (22 subjects) and who had at least one on-study tumor assessment using RECIST 1.1 (19 subjects). One subject withdrew consist before first on-study tumor assessment and two subjects died before first on-study tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GPX-150
Number analyzed (Participants) | 19
Participants | 3

2. Secondary Outcome: Number of Subjects Progression-free at Six Months Per RECIST 1.1
Description: This secondary efficacy endpoint is the progression-free rate (PFR) at 6 months, obtained from the Kaplan-Meier curve for progression-free survival (PFS).
Time Frame: 6 months from the beginning of the study treatment
Population: Consists of all subjects in the safety population who had at least one on-study tumor assessment using RECIST 1.1 (19 subjects). One subject withdrew consent before first on-study tumor assessment and two subjects died before first on-study tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GPX-150
Number analyzed (Participants) | 19
Participants | 8

3. Secondary Outcome: Number of Subjects Experiencing Adverse Events
Description: Subjects who received at least one dose were included in safety analyses. Adverse events were tabulated by System Organ Class (SOC) and Preferred Term (PT) and coded using MedDRA Version 19.1. Safety and tolerability was determined by frequency, nature, and severity of adverse events and the profile of toxicities.
Time Frame: From the beginning of study treatment and up to 12 months
Population: Subjects who received at least one dose of GPX-150 were included in the safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | GPX-150
Number analyzed (Participants) | 22
Participants | 22

4. Other Pre Specified Outcome: Number of Subjects With Tumor Response Per RECIST 1.1
Description: Tumor assessments using contrast enhanced computerized tomography (CT) scan of the Chest/Abdomen/Pelvis were performed to assess overall tumor burden. Response rate (RR), where response is defined as complete response (CR), partial response (PR), or stable disease (SD). Determination of CR or PR requires confirmation at the time of the next tumor assessment. An outcome of SD requires at least one assessment 6 weeks after the initiation of dosing. Progression is defined using RECIST 1.1, as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Assessed during screening, then every 6 weeks for the first 24 weeks on study, and then every 9 weeks for the next 24 weeks for up to 1 year. Subjects will be in the study for up to 1 year, or until disease progression or unacceptable toxicity.
Population: An on-study tumor assessment was done on 19 subjects within the ITT population; 2 subjects died before having a RECIST 1.1 measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | GPX-150
Number analyzed (Participants) | 19
Participants
  PD at final turmor assessment | 14
  SD at final tumor assessment | 5
  CR at final tumor assessment | 0
  PR at final tumor assessment | 0

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | GPX-150
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 22/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPX-150 (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Liposarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPX-150 (N=22)
Anemia (Blood and lymphatic system disorders) | 5 (12)
Abdominal pain (Gastrointestinal disorders) | 7 (10)
Constipation (Gastrointestinal disorders) | 10 (14)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (26)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (5)
Vomiting (Gastrointestinal disorders) | 10 (20)
Chest pain (General disorders) | 2 (3)
Chills (General disorders) | 3 (3)
Fatigue (General disorders) | 11 (17)
Oedema peripheral (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (4)
Hypersensitivity (Immune system disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Injection fraction decreased (Investigations) | 5 (7)
Anorexia nervosa (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Congenital, familial and genetic disorders) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No